CLINICAL TRIAL: NCT02179762
Title: Enhancing Active Surveillance With Exercise (EASE): A Pilot Randomized Trial in Localized Prostate Cancer Survivors
Brief Title: Vigorous or Moderate Exercise in Enhancing Active Surveillance in Patients With Localized Prostate Cancer
Acronym: EASE
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient staff
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE9814; NCI-2014-01313 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CASE9814 (Other: Case Comprehensive Cancer Center); P30CA043703 (NIH)
Record Dates: First submitted 2014-06-30; First posted 2014-07-02 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Recurrent Prostate Cancer; Stage I Prostate Cancer; Stage IIA Prostate Cancer; Stage IIB Prostate Cancer
Keywords: cancer survivor; prostate cancer; exercise; Active surveillance; EASE
MeSH Terms: conditions — Prostatic Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm I (moderate intensity exercise) (Experimental): Patients perform moderate intensity exercise on a stationary bike for 20-50 minutes, three days a week for 16 weeks.
  Interventions: Behavioral: moderate exercise intervention; Other: questionnaire administration; Other: laboratory biomarker analysis; Behavioral: Exercise Logs; Behavioral: Adherence; Behavioral: Exercise and body composition test
- Arm II (HIIT exercise on a standard stationary bike) (Experimental): Patients perform HIIT exercise on a standard stationary bike, three days a week for 16 weeks.
  Interventions: Behavioral: vigorous exercise intervention - standard; Other: questionnaire administration; Other: laboratory biomarker analysis; Behavioral: Exercise Logs; Behavioral: Adherence; Behavioral: Exercise and body composition test
- Arm III (HIIT exercise on a cybercycle) (Experimental): Patients perform HIIT exercise on a cybercycle using racing or other games, three days a week for 16 weeks.
  Interventions: Other: questionnaire administration; Other: laboratory biomarker analysis; Behavioral: vigorous exercise intervention - cybercycling; Behavioral: Exercise Logs; Behavioral: Adherence; Behavioral: Exercise and body composition test

INTERVENTIONS:
Behavioral: moderate exercise intervention — Perform moderate exercise therapy
  Arms: Arm I (moderate intensity exercise)
Behavioral: vigorous exercise intervention - standard — Perform HIIT exercise therapy on a standard stationary bike
  Arms: Arm II (HIIT exercise on a standard stationary bike)
Other: questionnaire administration — Ancillary studies: Functional Assessment of Cancer Therapy-General (FACT-G), Godin Leisure-Time Exercise questionnaire, 24-hour diet recalls, USDA 5 Step Multiple Pass Method, Memorial Anxiety Scale for Prostate Cancer, Pittsburgh Sleep Quality Index (PSQI)
Other: laboratory biomarker analysis — Correlative studies
Behavioral: vigorous exercise intervention - cybercycling — perform HIIT exercise on cybercycles aided by electronic racing and other games
  Arms: Arm III (HIIT exercise on a cybercycle)
Behavioral: Exercise Logs — The exercise physiologists will keep exercise logs and tracking sheets that log the date, start and stop time (duration) of exercise sessions as well as time in the THR and RPE for each exercise session.
Behavioral: Adherence — We will assess barriers to adhering to the exercise protocol by asking an open-ended question to solicit barriers. If the patient calls to cancel an exercise session, he will be called and probed for reasons
Behavioral: Exercise and body composition test — Height will be measured to the nearest 0.1 cm and weight will be measured to the nearest 0.1 kg. Waist and hip circumference will be measured to the nearest 1/8 inch. Whole body dual-energy X-ray absorptiometry scans will be conducted at baseline and end of treatment to quantify total body fat.

SUMMARY:
This randomized pilot clinical trial compares vigorous or moderate exercise in enhancing active surveillance in patients with prostate cancer that has not spread to nearby lymph nodes or to other parts of the body. Active surveillance involves watching the patient's condition but not giving any treatment unless test results show that the patient's condition is getting worse. Exercise may improve fitness, quality of life, brain health, and blood biomarkers in patients with prostate cancer on active surveillance. It is not yet known whether vigorous or moderate exercise works better in enhancing active surveillance in patients with localized prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the feasibility of performing vigorous intensity aerobic exercise using progressive, high-intensity interval training (HIIT) with standard stationary cycling and 'cybercycling' compared to moderate intensity aerobic exercise with standard stationary cycling in prostate cancer (PCa) survivors on active surveillance (AS).

II. To explore the potential effects of vigorous intensity aerobic exercise (HIIT) using standard cycling and 'cybercycling' compared to moderate intensity standard cycling on changes in quality of life (QoL), cognition, fitness circulating inflammatory biomarkers and PCa-specific markers of progression (prostate specific antigen [PSA], time to AT) in PCa survivors in active surveillance (AS); and, to explore if these effects may be mediated by changes in body fat.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients perform moderate intensity exercise on a stationary bike for 20-50 minutes, three days a week for 16 weeks.

ARM II: Patients perform HIIT exercise on a standard stationary bike, three days a week for 16 weeks.

ARM III: Patients perform HIIT exercise on a cybercycle using racing or other games, three days a week for 16 weeks.

After completion of study, patients are followed up at 6 and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Adult men of all races and body size with histologically confirmed localized PCa on AS
* Approved to be contacted by the treating urologist
* Meet screening criteria

  * Complete American Heart Association (AHA)/American College of Sports Medicine (ACSM) exercise questionnaire
  * Undergo cardiopulmonary exercise (CPX) testing utilizing a cycle ergometer. If the CPX test is terminated secondary to hemodynamic instability, arrhythmias or ischemic signs, the patient will be ineligible.

Exclusion Criteria:

* Patients unable to provide informed consent
* Patients participating in a structured exercise program in the past 6 months
* Patients not available for follow-up tests
* Patients with pre-existing medical conditions that would be a barrier to exercise

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-08-09 (Actual); Primary Completion 2018-07-23 (Actual); Study Completion 2018-07-23 (Actual)

PRIMARY OUTCOMES:
Overall attendance | Up to 16 weeks
  Average number of people who attend each session
Overall adherence to the exercise protocol as measured by average time in HIIT intervals for HIIT groups | Up to 16 weeks
  Average number of minutes in HIIT intervals which are defined as exercising at 80-90% WR_peak
Adherence to the exercise protocol as measured by average time in the target heart rate (THR) zone | Up to 16 weeks
  the target heart rate zone will be determined using the Karvonen formula: THR=((HRmax - HRrest) × % Intensity) + HRrest. Total time in this zone will be recorded every 5 minutes and the overall average will be recorded

SECONDARY OUTCOMES:
Average change in the Exercise Motivations Inventory (EMI-2) | Baseline up to 16 weeks
  The EMI-2 is a validated, 51 item instrument where each question is scored 0-5 and higher scores indicate greater motivation. Average changes will be analyzed using t-tests as well as mixed linear models adjusted for potential confounding factors.
Change in quality of life, measured using the Functional Assessment of Cancer Therapy (FACT) | Baseline up to 16 weeks
  A 25 item scale scored 0-4 where lower indicate greater quality of life. Paired t-tests will be used to evaluate change as well as mixed linear models adjusted for potential confounding factors.
Average change in fitness | Baseline up to 16 weeks
  Difference in VO2 maximum 30 second intake from beginning of study to end of treatment. Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in body mass index as a measure of body composition | Baseline up to 16 weeks
  Change in body mass index (function of height and weight) from baseline to end of treatment. Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in cognition | Baseline up to 16 weeks
  Average change in score of cognitive survey. Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in eating behaviors | Baseline up to 16 weeks
  61 items where higher scores indicate healthier eating behaviors. Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in leptin | Baseline up to 16 weeks
  Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in insulin | Baseline up to 16 weeks
  Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in adiponectin | Baseline up to 16 weeks
  Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in resistin | Baseline up to 16 weeks
  Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in IGF-1 | Baseline up to 16 weeks
  Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in IGFBP-1 | Baseline up to 16 weeks
  Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in IGFBP-3 | Baseline up to 16 weeks
  Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in TNF-alpha | Baseline up to 16 weeks
  Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Average change in the Exercise Causality Orientations Scale (ECOS) | Baseline up to 16 weeks
  The ECOS is a validated, 21 item instrument where each question is scored 1-7 and higher scores indicate greater motivation. Average changes will be analyzed using t-tests as well as mixed linear models adjusted for potential confounding factors.
Change in waist/hip circumference ratio as a measure of body composition | Baseline up to 16 weeks
  Change in waist and hip circumference ratio from baseline to end of treatment. Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.
Change in total body fat as a measure of body composition | Baseline up to 16 weeks
  Change in total body fat from baseline to end of treatment as measured by whole body dual-energy X-ray absorptiometry scans. Paired t-tests will be used to evaluate changes as well as mixed linear models adjusted for potential confounding factors.

CONTACTS AND LOCATIONS:
Overall Officials: Nora Nock, PhD, Principal Investigator — Case Comprehensive Cancer Center